CLINICAL TRIAL: NCT06961708
Title: A Phase 1, Randomized, Single-center, Double-blind, Placebo-controlled Study of Fosmanogepix Administered as Single and Multiple Doses in Healthy Adult Chinese Subjects
Brief Title: A Study of Fosmanogepix in Healthy Adult Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FMGX-CP-109
Expanded Access: NCT06433128 (Available)
Record Dates: First submitted 2025-04-24; First posted 2025-05-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Fosmanogepix; Manogepix; Chinese; Pharmacokinetics; Healthy adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (single dose) (Experimental): Participants will receive fosmanogepix or placebo by oral administration
  Interventions: Drug: Oral Fosmanogepix; Drug: oral placebo
- Cohort 2 (single dose) (Experimental): Participants will receive fosmanogepix or placebo by IV infusion
  Interventions: Drug: IV Fosmanogepix; Drug: IV placebo
- Cohort 3 (multiple dose) (Experimental): Participants will receive fosmanogepix or placebo as an IV infusion twice 12 hours apart on Day 1 followed by a maintenance daily dose of fosmanogepix or placebo via IV infusion from Day 2 to Day 7
  Interventions: Drug: IV Fosmanogepix; Drug: IV placebo
- Cohort 4 (multiple dose) (Experimental): The participants will receive fosmanogepix or placebo as an IV infusion twice 12 hours apart on Day 1 followed by an IV maintenance daily dose on Day 2 and Day 3, and then switched to oral administration (of fosmanogepix or placebo) daily from Day 4 to Day 7.
  Interventions: Drug: Oral Fosmanogepix; Drug: IV Fosmanogepix; Drug: IV placebo; Drug: oral placebo

INTERVENTIONS:
Drug: Oral Fosmanogepix — Oral Tablet
  Arms: Cohort 1 (single dose); Cohort 4 (multiple dose)
Drug: IV Fosmanogepix — IV infusion
  Arms: Cohort 2 (single dose); Cohort 3 (multiple dose); Cohort 4 (multiple dose)
Drug: IV placebo — Matching IV placebo
  Arms: Cohort 2 (single dose); Cohort 3 (multiple dose); Cohort 4 (multiple dose)
Drug: oral placebo — Matching oral placebo
  Arms: Cohort 1 (single dose); Cohort 4 (multiple dose)

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics and safety of the investigational drug fosmanogepix including its active moiety manogepix following a single dose and multiple doses (by intravenous infusion (IV) or orally) in healthy Chinese adults.

The study consists of 2 consecutive Parts (Part-1, single-dose part followed by Part-2, multiple-dose part) including a total of approximately 52 participants.

Part-1 duration will be up to 64 days including 4 visits at the clinical site and Part-2 duration will be up to 70 days including 5 visits at the clinical site. The study will include a total of 4 study sub-groups (Cohorts 1-4) in which fosmanogepix or placebo will be administered in different strengths orally or IV.

Participants will be enrolled and randomly assigned to study drug.

During the study, serial blood samples will be collected to understand how fosmanogepix is changed and eliminated from the body. Participants will also receive physical examination and other tests. This will help to understand if fosmanogepix is safe.

All data analyses will be descriptive (no statistical analysis will be provided).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 30.0 kg/m2 inclusive, and a total body weight > 45 kg for females and > 50 kg for males at Screening.
* Subjects who are overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, vital signs, creatinine, and estimated creatinine clearance (Cockcroft-Gault formula).

Exclusion Criteria:

* Active acute or chronic infection, including, but not limited to upper airway infection, urinary tract infection, or skin infection at Screening.
* Any condition possibly affecting drug absorption.
* Medical history of neurological disorders including abnormal movements or seizures.
* Use of prescription or non-prescription drugs, including vaccines, and dietary and herbal supplements from Screening or within five half-lives (whichever is longer) prior to the first dose of study drug and throughout the study.
* Screening supine blood pressure (BP) ≥ 140 mmHg (systolic) or ≥ 90 mmHg (diastolic), and pulse rate (PR) > 100 beats per minute (bpm) or < 50 bpm, following at least 5 minutes of supine rest.
* Body temperature higher than 37.5 °C.
* Screening supine 12 lead ECG demonstrating clinically relevant abnormalities that may affect subject safety or interpretation of study results.
* Subjects with any of the following abnormalities in clinical laboratory tests at Screening, as assessed by the local laboratory and confirmed by a single repeat test, if deemed necessary:
* AST or ALT ≥ 1.0 × ULN.
* Total bilirubin ≥ 1.5 × ULN.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of manogepix in Part-1 | pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, 240 hours postdose
Time to peak manogepix concentration (Tmax) of manogepix in Part-1 | pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, 240 hours postdose
Area under the plasma concentration vs. time curve for 0-24 hours (AUC24) of manogepix in Part-1 | pre-dose, 1, 2, 3, 4, 6, 8, 12, 24 hours postdose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of manogepix in Part-1 | pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, 240 hours postdose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of manogepix in Part-1 | pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, 240 hours postdose
Maximum Observed Plasma Concentration (Cmax) of manogepix in Part-2 | pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, 240, 360 hours postdose on Day 7
Time to peak manogepix concentration (Tmax) of manogepix in Part-2 | pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, 240, 360 hours postdose on Day 7
Area under the concentration-time curve at steady state over the dosing interval tau (AUCtau) of manogepix in Part-2 | pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, 240, 360 hours postdose on Day 7

SECONDARY OUTCOMES:
Number of participants reporting adverse events (AEs) in Part-1 | Screening to follow-up (Day 29-36)
Plasma protein binding of manogepix: Fraction unbound (fu) in Part 1 | pre-dose and 3 hours postdose
Number of participants reporting adverse events (AEs) in Part-2 | Screening to follow-up (Day 35-42)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Longchuan North Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-04-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT06961708/ICF_000.pdf